CLINICAL TRIAL: NCT00250094
Title: Clinical Benefit of Topoisomerase Downregulation: A Phase I Pilot Study
Brief Title: Clinical Benefit of Topoisomerase Downregulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0603C
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Ovarian Cancer
Keywords: Phase I; Ovarian Cancer; Ovary; Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — Topotecan; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topotecan and VP16 — Course 1A: On day 1 treatment will start with a continuous infusion of TPT at 0.4 mg/m2/day for 21 days. A pump will be used to deliver the TPT. The bag in the pump will be replaced every week for sterility precautions.
  Course 1B: On day 28, if ANC is >1,500 and platelets > 100,000, VP-16 will be administered orally at 50 mg/day for 14 days.

SUMMARY:
1.1 To determine the regulation of topoisomerase I and II following alternating prolonged exposure to topotecan and etoposide (VP-16)

1.2 To determine the time to progression and the objective response rate of this treatment in patients with incurable ovarian cancer.

DETAILED DESCRIPTION:
The rationale to study the downregulation of topoisomerase enzyme in ovarian cancer in relationship to the cell cycle distribution of the cancer cells after a prolonged continuous exposure to topo I and II poisons is to better understand the relationship between cell cycle and topo poisoning, which may lead to better clinical trial designs.

ELIGIBILITY:
Inclusion Criteria:

* All patients, 18 years of age or older, with incurable ovarian advanced cancer are eligible provided that they have measurable disease by CT-scan imaging, or evaluable disease by tumor markers, following the criteria described by Rustin et al. (14). (Response to a specific treatment has occurred if after two CA-125 samples there has been a 50% decrease, confirmed by a fourth sample (50% response), or a serial decrease over three samples of greater than 75% (75% response). The final sample has to be at least 28 days after the previous sample.)
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have a Zubrod performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of > 1,500 or cells/mm3 and platelet count >100,000/mm3 and absence of a regular red blood cell transfusion requirement.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine < 1.5 x upper limit of normal.

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded from this study.
* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-05; Primary Completion 2005-06 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To determine the regulation of topoisomerase I and II following alternating prolonged exposure to topotecan and etoposide (VP-16) | 3 years

SECONDARY OUTCOMES:
To determine the time to progression and the objective response rate of this treatment in patients with incurable ovarian cancer | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Claire F Verschraegen, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States